CLINICAL TRIAL: NCT04937166
Title: An Open-label Phase Ib Study of DSP107 for Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: A Study of Dual-SIgnaling Protein 107 (DSP107) for Patients With Hematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrolment
Sponsor: Kahr Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DSP107_002
Record Dates: First submitted 2021-06-06; First posted 2021-06-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: This study will involve sequential enrollment of approximately 36 patients accrued into six dose cohorts, each testing a different DSP107 dose level in combination with azacitidine (Part A) or DSP107 in combination with azacitidine and venetoclax (Part B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DSP107 in combination with azacitidine or azacitidine plus venetoclax. (Experimental): DSP107 will be administered by intravenous infusion once weekly during each 28-day cycle to all patients in this study.
  Azacitidine (75 mg/m2/day) will be administered subcutaneously or intravenously for the first 7 days of every cycle.
  Patients enrolled in Part B only will also receive venetoclax. During Cycle 1, venetoclax will be dose escalated daily to the goal dose of 400 mg daily. Patients will receive 100 mg on Day 1, 200 mg on Day 2 and 400 mg on Day 3 and onwards.
  Interventions: Biological: DSP107; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Biological: DSP107 — DSP107 (SIRPα - 4-1BBL) is a bi-functional, trimeric, fusion protein.
Drug: Azacitidine — Azacitidine is an analog of the pyrimidine nucleoside cytidine.
  Other Names: Vidaza
Drug: Venetoclax — Venetoclax is a B-cell lymphoma (BCL)-2 inhibitor
  Other Names: Venclexta, Venclyxto

SUMMARY:
This study will be divided into two parts, Parts A and B and will enroll patients with relapsed/refractory AML or MDS/chronic myelomonocytic leukemia (CMML) patients who have failed up to 2 prior therapeutic regimens.

Part A is a dose escalation study to explore the safety, efficacy, pharmacokinetic (PK) and pharmacodynamic (PD) profile of DSP107 when administered in combination with azacitidine (AZA).

Part B is a dose escalation study to explore the safety, efficacy, PK and PD profile of DSP107 when administered in combination with AZA and venetoclax (VEN).

DETAILED DESCRIPTION:
Part A is a dose escalation study in up to 4 cohorts of patients designed to test the safety and efficacy of DSP107 administered alone and in combination with AZA. The DSP107 starting dose level in Part A will be 0.3 mg/kg based on aggregate safety, PK and PD data from study DSP107_001, an ongoing study exploring the safety of escalating DSP107 doses in patients with advanced solid tumors. There will be a single DLT evaluation period, lasting 28 days, to determine the safety of DSP107 in combination with AZA. The safety, efficacy and PK data will be used to establish a recommended Phase II dose for potential future expansion cohorts and a starting dose for Part B.

Part B is a dose escalation study in 2 cohorts of patients that will test the safety and efficacy of DSP107 in combination with AZA and VEN. The starting dose for Part B will be at least one dose level lower than the DSP107 dose selected in Part A as being safe and effective in combination with AZA. Once a safe, effective dose has been established in Part B, a recommended phase 2 dose for patients with newly diagnosed AML will be agreed with the FDA at an End-of-Phase 1 meeting.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* White Blood Cell count < 20 x 10^9/L.
* Adequate organ function
* Relapsed/refractory AML or MDS/CMML patients who have failed up to 2 prior therapeutic regimens.

Exclusion Criteria:

* Acute Promyelocytic leukemia
* Symptomatic central nervous system (CNS) leukemia or patients with poorly controlled CNS leukemia
* Life-threatening (grade 4) immune-mediated adverse event related to prior immunotherapy
* Immune-mediated adverse reaction that required discontinuation of prior immunotherapy
* Past or current history of autoimmune disease or immune deficiency
* History of severe interstitial lung disease or severe pneumonitis or active pneumonitis
* Clinically significant and poorly compensated liver disease
* Prior organ allografts (such as renal transplant) requiring active immunosuppression
* Active graft versus host disease
* Treatment with systemic immunostimulatory within 4 weeks prior to initiation of study treatment
* Treatment with any CD47/SIRPα targeting agent or immune agonists
* Known allergy or hypersensitivity to any of the test compounds, materials or contraindication to test product
* Received live, attenuated vaccine within 4 weeks prior to first dose of study treatment
* Active Hepatitis B or C infection
* History or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease
* Pregnant or breast feeding or planning to become pregnant while enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Duration of the study, estimated to be 12 months
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Dose Limiting Toxicities (DLT) | At the end of Treatment Cycle 2 (within 2 months of treatment initiation)
  A DLT is defined as a clinically significant AE or laboratory abnormality that is related to DSP107 or the combination of DSP107 and AZA, but is unrelated to disease progression, intercurrent illness or concomitant medications
Response Rate (RR) including Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi) | Within 6 months of treatment initiation
  Response rates will be determined by assessing peripheral blood and bone marrow samples.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Within 6 months of treatment initiation
  Peripheral and bone marrow samples will be assessed to determine ORR. The ORR will measure the proportion of patients who achieve CR, CRi, complete remission with incomplete hematological recovery (CRh), complete remission with incomplete platelet recovery (CRp) or partial response (PR) within 6 months of treatment initiation, with or without cytogenetic response, hematological improvements and a morphologic leukemia-free state.
Morphologic Leukemia-Free (MLF) Rate | Within 6 months of treatment initiation
  Peripheral and bone marrow samples will be assessed to determine the proportion of patients who are morphologically leukemia-free within 6 months of treatment initiation.
Minimal Residual Disease (MRD) Status | Duration of the study, estimated to be 12 months
  Peripheral and bone marrow samples will be assessed to determine minimal residual disease (MRD) status at response and/or the best MRD response during study participation.
4-week Mortality Rate | Within 4 weeks of treatment initiation
  The proportion of patients who die within 4 weeks of treatment initiation.
DSP107 Serum Concentration | Duration of the study, estimated to be 12 months
  Serum samples will be collected to determine circulating levels of DSP107.
DSP107 anti-drug antibody (ADA) formation | Duration of the study, estimated to be 12 months
  Serum samples will be collected throughout the study for assessment of ADA formation using validated assay.
Change in Phenotypic and Activation Profiles of Peripheral Blood Mononuclear Cells | Duration of the study, estimated to be 12 months
  Whole blood samples will be collected throughout the study for immunophenotyping by flow cytometry and/or mass cytometry.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - The University of Texas MD Anderson Cancer Center, Department of Leukemia, Houston, Texas